CLINICAL TRIAL: NCT05626751
Title: A Multicenter, Open-label Extension Trial to Evaluate the Efficacy, Safety and Tolerability of HZN-825 in Patients With Diffuse Cutaneous Systemic Sclerosis
Brief Title: An Open-label Extension Trial of HZNP-HZN-825-301 in Adult Participants With Diffuse Cutaneous Systemic Sclerosis (Diffuse Cutaneous SSc)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was not stopped due to safety reasons
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HZNP-HZN-825-302; 2023-509783-23-00 (EU CTIS Number)
Record Dates: First submitted 2022-11-01; First posted 2022-11-25 (Actual); Results first posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-11

CONDITIONS: Diffuse Cutaneous Systemic Sclerosis; Sclerosis, Systemic
Keywords: Scleroderma; Forced vital capacity
MeSH Terms: conditions — Scleroderma, Diffuse; Scleroderma, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HZN-825 (Experimental): HZN-825 will be administered by mouth (PO) twice daily (BID) for 52 weeks
  Interventions: Drug: HZN-825

INTERVENTIONS:
Drug: HZN-825 — HZN-825 will be administered BID for 52 weeks

SUMMARY:
Primary Objectives:

1. The primary efficacy objective is to assess the efficacy of 52 weeks of open-label treatment with HZN-825 in participants with diffuse cutaneous systemic sclerosis, as measured by change from both baselines in forced vital capacity percent (FVC %) predicted.
2. The primary safety objective is to examine the safety and tolerability of 52 weeks of open-label treatment with HZN-825, inclusive of, but not limited to, adverse events (AEs), serious AEs (SAEs) and the adverse event of special interest (AESI), from Day 1 to 4 weeks after last dose.

DETAILED DESCRIPTION:
This is an open-label, repeat-dose, multicenter extension trial of HZNP-HZN-825-301. Participants who complete the double-blind Treatment Period (Week 52) in Trial HZNP-HZN-825-301 will be eligible to enter this 52-week extension trial. Participants entering this extension trial will complete the Week 52 Visit activities in HZNP-HZN-825-301 and will not complete the Safety Follow-up Visit 4 weeks after the last dose of trial drug in HZNP-HZN-825-301.

Acquired from Horizon in 2024.

ELIGIBILITY:
Key Inclusion Criteria:

1. Completed the double-blind Treatment Period (Week 52) in Trial HZNP-HZN-825-301; participants prematurely discontinued from trial drug in Trial HZNP-HZN-825-301 for reasons other than safety or toxicity can be included at the discretion of the Investigator after completing Trial HZNP-HZN-825-301 scheduled visits, including Week 52 assessments.

Key Exclusion Criteria:

1. Anticipated use of another investigational agent for any condition during the course of the trial.
2. New diagnosis of malignant condition after enrolling in Trial HZNP-HZN-825-301 (except successfully treated basal/squamous cell carcinoma of the skin or cervical cancer in situ).
3. Women of childbearing potential (WOCBP) or male participants not agreeing to use highly effective method(s) of birth control throughout the trial and for 4 weeks after last dose of trial drug as defined in the protocol.
4. Any new development with the participant's disease or condition or any significant laboratory test abnormality during the course of Trial HZNP-HZN-825-301 that, in the opinion of the Investigator, would potentially put the subject at unacceptable risk.
5. Pregnant or lactating women.
6. Participants will be ineligible if, in the opinion of the Investigator, they are unlikely to comply with the trial protocol or have a concomitant disease or condition that could interfere with the conduct of the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2022-11-04 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (65):
- United States (11):
  - Arizona Arthritis and Rheumatology Associates -4550 E Bell Rd, Phoenix, Arizona
  - UCLA Medical Center, Los Angeles, California
  - University of Miami Miller School of Medicine, Miami, Florida
  - IRIS Research and Development LLC, Plantation, Florida
  - DelRicht Clinical Research, LLC - Internal - Covington - PPDS, New Orleans, Louisiana
  - Boston University School Of Medicine, Boston, Massachusetts
  - Michigan Medicine University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic - Cancer Center - Rochester - PPDS, Rochester, Minnesota
  - Duke University Medical Center, Durham, North Carolina
  - Medical University of South Carolina (MUSC) - PPDS, Charleston, South Carolina
  - UT Physicians Rheumatology, Houston, Texas
- Argentina (8):
  - Framingham Centro Médico, La Plata, Buenos Aires
  - Consultorio Médico Dra. Rivera, Buenos Aires, Ciudad Autónoma de BuenosAires
  - Centro de Investigaciones Médicas Tucumán - PPDS, San Miguel de Tucumán, Tucumán Province
  - Centro de Investigaciones Reumatológicas, San Miguel de Tucumán, Tucumán Province
  - Clínica Mayo de U.M.C.B. S.R.L, San Miguel de Tucumán, Tucumán Province
  - Aprillus Asistencia e Investigacion de Arcis Salud SRL, Buenos Aires
  - Clínica Adventista Belgrano, Cuiudad Autónoma de Buenos Aires
  - I.R. Medical Center - Hospital de Dia, Mendoza
- Prosalud y Cia Ltda., Santiago, Región-MetropolitanadeSantiago, Chile
- Greece (3):
  - Laiko General Hospital of Athens, Athens, Attica
  - Euromedica Kianous Stavros, Thessaloniki
  - General Hospital of Thessaloniki ''Hippokratio'', Thessaloniki
- Israel (4):
  - The Chaim Sheba Medical Center - PPDS, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center Ichilov - PPDS, Tel Aviv, Tel Aviv
  - Rambam Health Care Campus - PPDS, Haifa
  - Rabin Medical Center - PPDS, Petah Tikva
- Azienda Sanitaria Universitaria Friuli Centrale - PO Universitario Santa Maria della Misericordia, Udine, Friuli Venezia Giulia, Italy
- Japan (7):
  - Hokkaido University Hospital, Sapporo, Hokkaidô
  - Sapporo Medical University Hospital, Sapporo, Hokkaidô
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - Saitama Medical University Hospital, Iruma-Gun, Saitama
  - Juntendo University Hospital, Bunkyo-Ku, Tokyo
  - Nippon Medical School Hospital, Bunkyo-Ku, Tokyo
  - Osaka Medical and Pharmaceutical University Hospital, Takatsuki-Shi, Ôsaka
- Mexico (8):
  - Centro de Estudios de Investigacion Basica Y Clinica SC, Guadalajara, Jalisco
  - Centro Integral Reumatologia SA de CV, Guadalajara, Jalisco
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, Mexico City
  - Centro de Investigación y Tratamiento Reumatológico S.C, San Miguel Chapultepec, Mexico City
  - Centro de Alta Especialidad En Reumatologia E Investigacion Del Potosi SC, Burócratas Del Estado, San Luis Potosí
  - Clinica de Investigacion en Reumatologia y Obesidad, Guadalajara
  - Unidad de Atencion Medica e Investigacion en Salud, Mérida
  - CITER, Centro de Investigacion y Tratamiento de las Enfermedades Reumaticas SA de CV, México
- Poland (4):
  - Malopolskie Centrum Kliniczne, Krakow, Lesser Poland Voivodeship
  - Twoja Przychodnia NCM, Nowa Sól, Lubusz Voivodeship
  - Medicover Integrated Clinical Services sp. z o.o - MICS - PPDS, Warsaw, Masovian Voivodeship
  - Centrum Medyczne Reuma Park NZOZ, Warsaw, Masovian Voivodeship
- Hospital de Santa Maria-Avenida Prof. Egas Moniz - PPDS, Lisbon, Portugal
- Romania (3):
  - Sf.Maria Clinical Hospital, Bucharest, București
  - Dr I Cantacuzino Clinical Hospital, Bucharest, București
  - Centrul Medical de Diagnostic si Tratament Ambulator NEOMED SRL, Brasov
- Serbia (2):
  - Institute of Rheumatology - PPDS, Belgrade
  - Institute for Treatment and Rehabilitation Niska Banja, Niška Banja
- South Korea (4):
  - Chonnam National University Hospital, Gwangju, Gwangju Gwang'yeogsi
  - Seoul National University Bundang Hospital, Seongnam, Gyeonggido
  - Hanyang University Seoul Hospital, Seongdong-gu, Seoul Teugbyeolsi
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
- Spain (7):
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario A Coruña, A Coruña
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Hospital de La Santa Creu i Sant Pau, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Quironsalud Infanta Luisa, Seville
  - Hospital Universitario Doctor Peset, Valencia
- Royal Free Hospital, London, London, City of, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 77 research centers in Argentina, Austria, Chile, France, Germany, Greece, Israel, Italy, Japan, South Korea, Mexico, Poland, Portugal, Romania, Serbia, Spain, Switzerland, the United Kingdom, and the United States between November 2022 to February 2025.
Pre-assignment Details: This trial is an open-label extension (OLE) of the parent trial HZNP-HZN-825-301, in which participants received either HZN-825 300 mg twice daily (BID), HZN-825 300 mg once daily (QD), or placebo. Participants in this OLE trial all received the same dose regimen: open-label HZN-825 300 mg BID, orally, for 52 weeks. Participants are analyzed according to the group determined by the treatment received in the parent trial.
Groups:
- HZN-825 300 mg QD in Parent Trial: Participants who received HZN-825 300 mg QD in the parent trial received HZN-825 300 mg orally BID in this OLE extension for 52 weeks.
- HZN-825 300 mg BID in Parent Trial: Participants who received HZN-825 300 mg BID in parent trial continued to receive HZN-825 300 mg orally BID in this OLE extension for 52 weeks.
- Placebo in Parent Trial: Participants who received Placebo in parent trial received HZN-825 300 mg orally BID in this OLE extension for 52 weeks.
Period: Overall Study
Arm/Group | HZN-825 300 mg QD in Parent Trial | HZN-825 300 mg BID in Parent Trial | Placebo in Parent Trial
Started | 62 | 52 | 60
Full Analysis Set | 62 | 52 | 60
Safety Analysis Set (Participants in the safety analysis set are analyzed based on the treatment received, not on the groups to which they were randomized. This analysis set was analyzed according to the treatment actually received.) | 62 | 53 | 59
Completed | 15 | 15 | 17
Not Completed | 47 | 37 | 43
Not completed — Lost to Follow-up | 1 | 2 | 1
Not completed — Trial Terminated by Sponsor | 39 | 30 | 37
Not completed — Withdrawal by Subject | 7 | 5 | 5

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) included all participants who were enrolled and received at least one full or partial dose of HZN-825 in this extension trial. Participants in this analysis set were analyzed according to the group determined by the treatment that the participant received in the parent trial HZNP-HZN-825-301.
Groups:
- Total: Total of all reporting groups
Arm/Group | HZN-825 300 mg QD in Parent Trial | HZN-825 300 mg BID in Parent Trial | Placebo in Parent Trial | Total
Number analyzed (Participants) | 62 | 52 | 60 | 174
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (12.7) | 49.8 (11.2) | 48.5 (12.4) | 49.0 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 44 | 50 | 140
  Male | 16 | 8 | 10 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 20 | 25 | 71
  Not Hispanic or Latino | 36 | 32 | 35 | 103
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 2
  Asian | 5 | 7 | 9 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 2
  Black or African American | 2 | 1 | 2 | 5
  White | 54 | 36 | 44 | 134
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 6 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Forced Vital Capacity Percentage (FVC%) Predicted at Week 52
Description: FVC is the amount of air that can be forcibly exhaled from the lungs after taking the deepest breath possible, as measured by spirometry. FVC is a measure of respiratory function. FVC% predicted was calculated by taking the observed FVC measurement and dividing it by a predicted value multiplied by 100 (% FVC predicted = (FVC observed/FVC predicted) x 100). The predicted value is an average of the normal FVC volume for a person of the same sex, ethnicity, age and height.
Time Frame: Baseline and Week 52
Population: The FAS included all participants who were enrolled and received at least one full or partial dose of HZN-825 in this extension trial. Only participants with available data were included in this endpoint. Participants were analyzed according to the group determined by the treatment that the participant received in the parent trial HZNP-HZN-825-301.
Measure: Mean (Standard Deviation); unit: % predicted FVC
Arm/Group | HZN-825 300 mg QD in Parent Trial | HZN-825 300 mg BID in Parent Trial | Placebo in Parent Trial
Number analyzed (Participants) | 14 | 15 | 13
% predicted FVC | -1.36 (8.46) | -7.95 (15.36) | -0.82 (4.09)

2. Primary Outcome: Number of Participants Who Experienced Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event (AE) was defined as any untoward medical occurrence in a trial participant who received an investigational product (IP), regardless of a causal relationship with treatment. An AE could be any unfavorable and unintended sign (including abnormal laboratory findings), symptom, or disease temporally associated with the use of an IP. TEAEs were defined as events that began or worsened in severity on or after the first dose of treatment through 28 days after the last dose or the cutoff date for ongoing participants. Serious TEAEs were those that resulted in death, were life-threatening, required or prolonged hospitalization, caused significant disability/incapacity, led to a congenital anomaly/birth defect, or were considered other important medical events. Clinically significant changes in vital signs, electrocardiograms (ECGs), and laboratory tests were included as TEAEs.
Time Frame: From 1st dose to last dose + 28 days; median (min, max) time on trial was 8.5 (1.0, 14.0) months
Population: The safety analysis set (SAS) included all participants who had received at least one dose or partial dose of HZN-825 in the extension trial.
Measure: Count of Participants; unit: Participants
Arm/Group | HZN-825 300 mg QD in Parent Trial | HZN-825 300 mg BID in Parent Trial | Placebo in Parent Trial
Number analyzed (Participants) | 62 | 53 | 59
Participants
  TEAEs | 34 | 37 | 35
  Serious TEAEs | 2 | 2 | 5

3. Primary Outcome: Number of Participants Who Experienced AEs of Special Interest (AESI)
Description: The following AESI was identified for this trial: Orthostatic hypotension defined as a reduction of systolic blood pressure by ≥20 mmHg or reduction of diastolic blood pressure by ≥10 mmHg and associated with symptoms such as lightheadedness, blurred vision, weakness, fatigue, cognitive impairment, nausea, palpitations, tremulousness, headache, presyncope or syncope.
Time Frame: Day 1 and at Weeks 4, 28 and 52
Population: The SAS included all participants who had received at least one dose or partial dose of HZN-825 in the extension trial.
Measure: Count of Participants; unit: Participants
Arm/Group | HZN-825 300 mg QD in Parent Trial | HZN-825 300 mg BID in Parent Trial | Placebo in Parent Trial
Number analyzed (Participants) | 62 | 53 | 59
Participants | 0 | 0 | 0

4. Primary Outcome: Number of Participants Using Any Concomitant Medication
Description: Concomitant medications were defined as any medication that was ongoing, had a start date on or after the first dose of the trial drug, or had a stop date on or after the first dose date.
Time Frame: From 1st dose to last dose + 28 days; median (min, max) time on trial was 8.5 (1.0, 14.0) months
Population: The SAS included all participants who had received at least one dose or partial dose of HZN-825 in the extension trial.
Measure: Count of Participants; unit: Participants
Arm/Group | HZN-825 300 mg QD in Parent Trial | HZN-825 300 mg BID in Parent Trial | Placebo in Parent Trial
Number analyzed (Participants) | 62 | 53 | 59
Participants | 62 | 52 | 58

ADVERSE EVENTS:
Time Frame: All-cause mortality: from enrollment to end of trial; median (min, max) time on trial 9.0 (0.8, 15.2) months. AEs: from 1st dose to last dose + 28 days; median (min, max) time on trial was 8.5 (1.0, 14.0) months.
Description: All-cause mortality is reported for all participants enrolled in the trial. Serious adverse events and other adverse events are reported for all participants who received at least one dose of IP.
Arm/Group | HZN-825 300 mg QD in Parent Trial | HZN-825 300 mg BID in Parent Trial | Placebo in Parent Trial
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/52 | 0/60
Serious Adverse Events (participants affected / at risk) | 2/62 | 2/53 | 5/59
Other Adverse Events (participants affected / at risk) | 17/62 | 18/53 | 20/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HZN-825 300 mg QD in Parent Trial (N=62) | HZN-825 300 mg BID in Parent Trial (N=53) | Placebo in Parent Trial (N=59)
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Dengue fever (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Extremity necrosis (Vascular disorders) | 0 | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HZN-825 300 mg QD in Parent Trial (N=62) | HZN-825 300 mg BID in Parent Trial (N=53) | Placebo in Parent Trial (N=59)
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 5
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 2 | 3
Nausea (Gastrointestinal disorders) | 1 | 1 | 3
Vomiting (Gastrointestinal disorders) | 3 | 3 | 0
COVID-19 (Infections and infestations) | 3 | 4 | 2
Nasopharyngitis (Infections and infestations) | 3 | 4 | 5
Pharyngitis (Infections and infestations) | 0 | 3 | 0
Urinary tract infection (Infections and infestations) | 3 | 3 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 | 0 | 3
Hypotension (Vascular disorders) | 4 | 0 | 0

LIMITATIONS AND CAVEATS:
The trial was terminated early as the parent trial (HZNP-HZN-325-301) was terminated due to meeting pre-defined criteria for futility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2024-10-14): https://cdn.clinicaltrials.gov/large-docs/51/NCT05626751/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-11): https://cdn.clinicaltrials.gov/large-docs/51/NCT05626751/SAP_001.pdf